CLINICAL TRIAL: NCT01667770
Title: Dural Graft Equivalent Comparison Trial
Acronym: DECOMPRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11BN113
Record Dates: First submitted 2012-08-14; First posted 2012-08-17 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Chiari Malformation
MeSH Terms: conditions — Arnold-Chiari Malformation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- surgery - autologous graft (Active Comparator): surgical intervention: decompression of Chiari malformation by suboccipital craniectomy using autologous graft
  Interventions: Procedure: decompression of Chiari malformation
- surgery - non-autologous graft (Active Comparator): surgical intervention: decompression of Chiari malformation by suboccipital craniectomy using using non-autologous graft
  Interventions: Procedure: decompression of Chiari malformation

INTERVENTIONS:
Procedure: decompression of Chiari malformation — Removal of a small section of bone at the back of the skull (posterior foramen magnum decompression) or upper cervical spine. During surgery, the covering of the brain (dura) is enlarged with a graft (autologous or non-autologous).

SUMMARY:
This research study is to find out which types of dural grafts used during surgery for Chiari Malformations are superior. We believe that autologous dural grafts are superior to non-autologous grafts.

DETAILED DESCRIPTION:
The study compares autologous grafts vs. non-autologous grafts. Non-autologous grafts include synthetics and grafts from animals. Autologous grafts have a better side-effect profile than non-autologous grafts. We believe this improved side-effect profile will result in a decreased incidence of reoperation for post-operative infections and post-operative fluid collections (pseudomeningoceles and seromas). Study is open to all non-pregnant minor and adult subjects. Subjects must have symptomatic Chiari Malformation described as > or equal to 6mm descent of the cerebellar tonsils below the foramen magnum with accompanying headaches and/or neurologic findings (arm pain/weakness, myelopathy, etc.). After the 12-month follow-up is completed on the first 100 subjects there will be an interim analysis of the results in order to determine whether one of the treatments has a statistically superior outcome. If a statistically superior outcome is noted, the trial will stop after being reviewed by a data monitoring committee. If no statistically significant difference is seen at one year, the study will continue until the 12-month follow-up is completed on the 200th patient.

ELIGIBILITY:
Inclusion Criteria:

* Minor or adult males and females
* Symptomatic Chiari Malformation
* Greater or equal to 6mm descent of the cerebellar tonsils below the foramen magnum
* Headaches and/or neurologic findings (e.g., arm pain/weakness, myelopathy, etc.)

Exclusion Criteria:

* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-01-18 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Complications encountered during the subject's post-operative care | 2 years
  After the 12-month follow-up is completed on the first 100 subjects there will be an interim analysis of the results in order to determine whether one of the treatments has a statistically superior outcome. If a statistically superior outcome is noted, the trial will stop after being reviewed by a data monitoring committee. If no statistically significant difference is seen at one year, the study will continue until the 12-month follow-up is completed on the 200th patient.

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Spetzler, M.D., Principal Investigator — Barrow Neurosurgical Associates
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States